CLINICAL TRIAL: NCT06718686
Title: Rifaximin in Dementia Trial (RIDE): Gut-Brain Modulation With Rifaximin SSD in Dementia
Brief Title: Rifaximin SSD in Dementia Trial
Acronym: RIDE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jasmohan Bajaj (U.S. Federal Agency)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Jasmohan Bajaj, Staff Physician, Hunter Holmes Mcguire Veteran Affairs Medical Center
Organization: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Allocation: Not Applicable | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 1817324
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Dementia Alzheimer Type; Dementia Associated With Cerebrovascular Disease
Keywords: dementia; rifaximin; gut-brain; Alzheimer's; vascular dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia; Dementia, Vascular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Patients will be given placebo and actual drug sequentially with the order hidden
  Interventions: Drug: Placebo
- Rifaximin SSD 40mg IR BID (Experimental): Patients will be given placebo and actual drug sequentially with the order hidden
  Interventions: Drug: Rifaximin SSD 40 mg IR tablet

INTERVENTIONS:
Drug: Rifaximin SSD 40 mg IR tablet — Drug therapy vs placebo
  Arms: Rifaximin SSD 40mg IR BID
Drug: Placebo — Placebo drug
  Arms: Placebo

SUMMARY:
Using a new formulation of rifaximin, a non-absorbable antibiotic, to test if it can affect microbes in the gut of patients with dementia favorably.

DETAILED DESCRIPTION:
Hypothesis: Rifaximin SSD therapy is safe and well tolerated in patients with AD and VaD with beneficial changes in systemic inflammation and systemic biomarkers of dementia due to improvement in microbiota function compared to placebo-related changes in a single-blind, placebo-controlled Phase 1b/2a trial .

Overall Objective: In a single blind placebo-controlled trial in patients with Alzheimer's or vascular dementia, to determine the effect of rifaximin SSD compared to placebo on gut microbial structure and function, cognitive and daily function, and caregiver burden.

ELIGIBILITY:
Inclusion Criteria:

* Probable Alzheimer's Disease (AD) or Vascular Dementia (VaD) mild or moderate based on Clinical Dementia Rating Scale.
* Males and Females Age ≥ 65 years
* Community living with availability of caregiver to accompany participant to study visits and to participate in the study.
* Able to consent or legal guardian who can consent (with participant assent).
* Legally authorized representative (LAR) and caregiver for the study is the same individual.
* Fluency (both participant and caregiver) in written and spoken English to participate in study visits.

Exclusion Criteria:

* Dementia not due to AD or VaD
* Clinically significant agitation or aggression (requiring treatment with antipsychotic medication)
* Delusions and/or hallucinations
* Severe psychopathology including major depression
* Unstable, severe, or poorly controlled medical conditions evident from physical examination or clinical history
* Visual and/or hearing disorder that prevents completion of neuropsychologic evaluations.
* Diarrhea
* Hypersensitivity to rifaximin, components of rifaximin,
* and any rifamycin antimicrobial agent
* Antibiotic use in the prior 6 months
* Taking medications that interact with Rifaximin. P-glycoprotein (P-gp) inhibitor treatment is permitted as long as the use of P-gp inhibitors is discussed with the investigator.
* History of alcohol and/or drug abuse
* Participation in another investigational drug trial in the last 30 days

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in stool and serum short-chain fatty acid levels | 10 weeks
  Change in SCFA in stool and serum in rifaximin SSD phase vs placebo phase
Change in bile acids in stool and serum | 10 weeks
  Change in bile acids in stool and serum in rifaximin SSD phase vs placebo phase

SECONDARY OUTCOMES:
Systemic inflammatory change | 10 weeks
  serum lipopolysaccharide-binding protein (LBP), inflammatory cytokines (IL-6, TNF-α, IL-10, IL-1β) in placebo phase vs Rifaximin SSD phase
Stool microbiome composition | 10 weeks
  16SrRNA microbiome composition and diversity change in placebo vs Rifaximin SSD phase
Change in dementia biomarkers | 10 weeks
  Plasma concentrations of Aβ42 and Aβ40 to calculate amyloid-β (Aβ)42/40 ratio and plasma concentration of phospho-tau (p-tau)181 in placebo vs Rifaximin SSD phase
MMSE | 10 weeks
  Change in MMSE between the 2 phases
Cognitive testing using Psychometric Hepatic Encephalopathy Score | 10 weeks
  Change in PHES in placebo vs rifaximin SSD phase
Clinical Dementia Rating - Sum of Boxes (CDR-SB) | 10 weeks
  Change in CDR-SB in placebo vs Rifaximin SSD phase
EncephalApp Stroop performance | 10 weeks
  Change in off time and on time in seconds between placebo and rifaximin SSD phases
Critical flicker fusion analysis | 10 weeks
  change in threshold to see CFF fusion in rifaximin SSD vs placebo phases
Katz Index of Independence in Activity of Daily Living (ADL) | 10 weeks
  change in the score above judged by caregivers in placebo vs Rifaximin SSD phase
Lawton-Brody Instrumental Activities of Daily Living (IADL) | 10 weeks
  Change in instrument score above by caregivers in rifaximin SSD vs placebo phase
Zarit Burden Interview short form | 10 weeks
  Change in instrument score above by caregivers in rifaximin SSD vs placebo phase
Sickness Impact profile | 10 weeks
  change in score of the QOL instrument above in placebo vs rifaximin SSD phases
PROMIS-29 | 10 weeks
  change in score of the QOL instrument above in placebo vs rifaximin SSD phases
Safety | 10 weeks
  Serious adverse event rates in placebo versus rifaximin SSD phases

CONTACTS AND LOCATIONS:
Overall Officials: Jasmohan Bajaj, Principal Investigator — Richmond VA Medical Center
Locations (1):
- Richmond VA Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Not IRB approved to do so